CLINICAL TRIAL: NCT02351440
Title: Effect of Preoperative Duloxetine on Quality of Recovery After Outpatient Laparoscopic Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Meghan Rodes, Assistant Professor, Department of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00096889
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Quality of Recovery; Gynecologic Surgery; Laparoscopy
Keywords: duloxetine
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): duloxetine 60mg PO
  Interventions: Drug: duloxetine
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: duloxetine — patients will be randomized to receive either duloxetine or placebo
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to determine the effect of preoperative duloxetine on postoperative quality of recovery after ambulatory surgery, specifically laparoscopic gynecological surgery.

DETAILED DESCRIPTION:
It has been demonstrated that female patients have poor quality of surgical recovery compared to male patients.1 Increased sensitivity to pain and increased susceptibility to postoperative nausea and vomiting have been attributed as causal factors.2, 3 Currently, few strategies have been shown to improve quality of recovery in female patients undergoing laparoscopic hysterectomy.4 A better recovery in female patients undergoing outpatient laparoscopy is particularly desirable since those patients do not have access to potent intravenous medications and nursing support after hospital discharge.

In addition, pain after ambulatory surgery remains an unsolved problem in The United States and Europe.5,6 It is associated with delayed hospital discharge and it can result to an increased opioid consumption with adverse side effects. The concept of multimodal analgesic technique was introduced more than 15 years ago and several techniques have been studied over the years including NSAIDs, acetaminophen, membrane stabilizers, ketamine, and local and regional anesthetic techniques.7,8 Both serotonin and norepinephrine have involvement in modulation of pain mechanisms in the central nervous system. Duloxetine is a selective serotonin and norepinephrine reuptake inhibitor that has been used for mitigation of pain in such conditions as chronic musculoskeletal pain, diabetic peripheral neuropathic pain, post-herpetic neuralgia, and fibromyalgia.9,10 Duloxetine was also found to reduce postoperative morphine requirements in patients undergoing knee replacement surgery.11 The MQOR 40 is a validated instrument that was specifically design to evaluate patient recovery after anesthesia and surgery.12 This instrument can be particularly valid to examine interventions which affect different spheres of patient recovery as is the case of duloxetine.

A suicidal behavior questionnaire (SBQ-R) will be used to screen for suicidal risk among potential subjects. If any subject exhibits suicidal ideation as a result of scoring high on the questionnaire, there surgeon and/or primary care provider will be notified by the principal investigator.

The objective of this study is to determine the effect of preoperative duloxetine on postoperative quality of recovery after ambulatory surgery.

Significance: Use of preoperative duloxetine may improve patient's quality of recovery, decrease postoperative pain, opioid consumption and opioid related side effects after ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* outpatient gynecological laparoscopy
* ASA PS 1 and 2
* fluent in English

Exclusion Criteria:

* history of allergy to duloxetine, history of chronic opioid use, pregnant patients, preoperative SSRI or SNRI use, prolonged QT interval on ECG

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
QOR-40 global score | 24 hours

SECONDARY OUTCOMES:
intraoperative opioid consumption | 1 hour
  measure intraoperative opioid consumption in morphine IV equivalents in mg

CONTACTS AND LOCATIONS:
Locations (1):
- Prentice Womens Hospital, Chicago, Illinois, United States